CLINICAL TRIAL: NCT01932801
Title: Harm Reduction With Pharmacotherapy for Homeless Adults With Alcohol Dependence
Brief Title: Harm Reduction With Pharmacotherapy (HaRP)
Acronym: HaRP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Alkermes, Inc. (Industry)
Responsible Party: Principal Investigator, Susan Collins, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 45134; 1R01AA022309-01 (NIH)
Record Dates: First submitted 2013-08-22; First posted 2013-08-30 (Estimated); Results first posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Use Disorder
Keywords: harm reduction, naltrexone, alcohol use disorder, homelessness
MeSH Terms: conditions — Alcoholism; Harm Reduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking of the double-blind portion of the study was quadruple until after all data had been collected, when they were unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Assessment-only (No Intervention): Assessment-only control condition
- HRC (Active Comparator): Harm reduction counseling, which entails provision of feedback and support of harm reduction goals and safer drinking provided at one-month intervals over a 3-month period.
  Interventions: Behavioral: HRC
- XR-NTX+HRC (Experimental): 3 doses of active medication (380 mg injection/month) + Harm reduction counseling at one-month intervals over three months.
  Interventions: Drug: XR-NTX; Behavioral: HRC
- Placebo+HRC (Placebo Comparator): 3 doses of placebo + harm reduction counseling at one-month intervals over a three-month period
  Interventions: Other: Placebo; Behavioral: HRC

INTERVENTIONS:
Drug: XR-NTX
  Arms: XR-NTX+HRC
Other: Placebo
  Arms: Placebo+HRC
Behavioral: HRC
  Arms: HRC; Placebo+HRC; XR-NTX+HRC

SUMMARY:
The goal of this study is to test the efficacy of extended-release naltrexone and harm reduction counseling in reducing alcohol-related harm among homeless people with alcohol dependence.

DETAILED DESCRIPTION:
Homelessness and alcohol dependence are commonly co-occurring and serious public health issues. Unfortunately, abstinence-based alcohol treatment approaches are minimally effective in engaging and successfully treating homeless individuals with alcohol dependence. There have therefore been calls for more flexible and client-centered approaches tailored to this population's needs. Innovative, low-barrier approaches (e.g., Housing First and alcohol management programs) have been applied with this population and are efficacious in reducing alcohol use and related problems as well as utilization of publicly funded services and associated costs. Such approaches have been referred to as harm-reduction interventions because they focus on reducing alcohol-related harm for affected individuals and their communities without requiring a commitment to abstinence-based goals. Although psychosocial, harm-reduction approaches are beginning to proliferate for this population, there are few pharmacological counterparts to support and enhance these efforts. One medication that could address this treatment gap is extended-release naltrexone (XR-NTX; marketed as Vivitrol®). XR-NTX is a 30-day, extended release formulation of the opioid receptor antagonist, naltrexone, and is administered monthly via gluteal intramuscular injection. The proposed Phase II study features a four-arm RCT (N=300) designed to test the efficacy of XR-NTX as a pharmacological adjunct to existing psychosocial harm-reduction services provided by community agencies to homeless people with alcohol dependence. The proposed study will include a 24-week follow-up and will test the relative efficacy of 3 active treatment combinations-1) XR-NTX+harm reduction counseling, 2) placebo+harm reduction counseling and 3) harm reduction counseling only (HRC)-compared to the services as usual (TAU) that all participants receive from community agencies. This proposed design will allow us to dismantle active treatment components and thereby detect potential "placebo effects" of both the administration of an injection and attention from a medical professional. In this study, there are three primary specific aims. First, we will test the relative efficacy of XR-NTX, placebo and HRC compared to TAU in decreasing alcohol quantity, frequency and alcohol-related problems. Second, we will test hypothesized mediators of the intervention effects. Specifically, we hypothesize that the active treatments will precipitate increases in motivation to change and decreases in craving, which, in turn, will mediate the active treatment effects on alcohol outcomes. Finally, we will test treatment effects on publicly funded service costs (i.e., emergency medical services, ER visits, hospital admissions, and county jail). It is hypothesized that XR-NTX, placebo and HRC groups will show greater decreases in publicly funded service costs than the TAU group.

ELIGIBILITY:
Inclusion Criteria:

* being a registered client at one of the named partnering sites
* being at least 21 years of age (for legal reasons)
* agreeing to use an adequate form of birth control (if female and in childbearing years) fulfilling criteria for current alcohol dependence according to DSM-IV-TR criteria as determined by the SCID-I/P

Exclusion Criteria:

* refusal or inability to consent to participation in research
* constituting a risk to safety and security of other clients or staff
* known sensitivity or allergy to naltrexone/XR-NTX
* current treatment with naltrexone/XR-NTX
* being pregnant or nursing
* suicide attempts within the past year
* renal insufficiency/serum creatinine level > 1.5
* current opioid dependence according to the DSM-IV-TR criteria
* liver transaminases (AST, ALT) > 5 times the upper limit of normal (ULN)
* clinical diagnosis of decompensated liver disease

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Collins, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington - Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Collins SE, Saxon AJ, Duncan MH, Smart BF, Merrill JO, Malone DK, Jackson TR, Clifasefi SL, Joesch J, Ries RK. Harm reduction with pharmacotherapy for homeless people with alcohol dependence: protocol for a randomized controlled trial. Contemp Clin Trials. 2014 Jul;38(2):221-34. doi: 10.1016/j.cct.2014.05.008. Epub 2014 May 17. PMID 24846619
- [Background] Collins SE, Duncan MH, Saxon AJ, Taylor EM, Mayberry N, Merrill JO, Hoffmann GE, Clifasefi SL, Ries RK. Combining behavioral harm-reduction treatment and extended-release naltrexone for people experiencing homelessness and alcohol use disorder in the USA: a randomised clinical trial. Lancet Psychiatry. 2021 Apr;8(4):287-300. doi: 10.1016/S2215-0366(20)30489-2. Epub 2021 Mar 10. PMID 33713622
- [Background] Fentress TSP, Wald S, Brah A, Leemon G, Reyes R, Alkhamees F, Kramer M, Taylor EM, Wildhood M, Frohe T, Duncan MH, Clifasefi SL, Collins SE. Dual study describing patient-driven harm reduction goal-setting among people experiencing homelessness and alcohol use disorder. Exp Clin Psychopharmacol. 2021 Jun;29(3):261-271. doi: 10.1037/pha0000470. PMID 34264737
- [Background] Goldstein SC, Spillane NS, Tate MC, Nelson LA, Collins SE. Measurement invariance and other psychometric properties of the Short Inventory of Problems (SIP-2R) across racial groups in adults experiencing homelessness and alcohol use disorder. Psychol Addict Behav. 2023 Mar;37(2):199-208. doi: 10.1037/adb0000833. Epub 2022 May 5. PMID 35511527

RESULTS

PARTICIPANT FLOW:
Groups:
- XR-NTX+HRC: 3 doses of active medication (380 mg injection/month) + Harm reduction counseling at one-month intervals over three months.
  XR-NTX+HRC
- Placebo+HRC: 3 doses of placebo + harm reduction counseling at one-month intervals over a three-month period
  Placebo+HRC
- Harm-reduction Counseling (HRC): Harm reduction counseling, which entails provision of feedback and support of harm reduction goals and safer drinking provided at one-month intervals over a 3-month period.
  HRC
Period: Overall Study
Arm/Group | XR-NTX+HRC | Placebo+HRC | Harm-reduction Counseling (HRC) | Assessment-only
Started | 74 | 78 | 79 | 77
Week 0 Session | 67 | 66 | 71 | 65
Week 4 Session | 54 | 54 | 60 | 41
Week 8 Session | 51 | 48 | 56 | 42
Week 12 Session | 56 | 50 | 55 | 40
Week 24 Session | 49 | 46 | 53 | 40
Week 36 Session | 48 | 48 | 54 | 40
Completed | 48 | 48 | 54 | 40
Not Completed | 26 | 30 | 25 | 37

BASELINE CHARACTERISTICS:
Groups:
- HRC - Harm Reduction Counseling: Harm reduction counseling, which entails provision of feedback and support of harm reduction goals and safer drinking provided at one-month intervals over a 3-month period.
  HRC
- Total: Total of all reporting groups
Arm/Group | Assessment-only | HRC - Harm Reduction Counseling | XR-NTX+HRC | Placebo+HRC | Total
Number analyzed (Participants) | 77 | 79 | 74 | 78 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.51 (9.50) | 49.38 (7.35) | 49.27 (9.11) | 46.55 (10.46) | 48.17 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 11 | 10 | 50
  Male | 61 | 66 | 63 | 68 | 258
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 6 | 7 | 34
  Not Hispanic or Latino | 67 | 67 | 68 | 71 | 273
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 13 | 11 | 8 | 50
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 1 | 3
  Black or African American | 16 | 24 | 33 | 28 | 101
  White | 28 | 24 | 20 | 24 | 96
  More than one race | 14 | 10 | 8 | 13 | 45
  Unknown or Not Reported | 0 | 8 | 1 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Quantity
Description: Using the Alcohol Quantity and Use Assessment, we will collect data on peak alcohol quantity.
Time Frame: Baseline, week 4, week 8, week 12, week 24, week 36
Measure: Mean (Standard Deviation); unit: number of drinks on peak occasion
Groups:
- HRC (Harm Reduction Counseling): Harm reduction counseling, which entails provision of feedback and support of harm reduction goals and safer drinking provided at one-month intervals over a 3-month period.
  HRC
Arm/Group | Assessment-only | HRC (Harm Reduction Counseling) | XR-NTX+HRC | Placebo+HRC
Number analyzed (Participants) | 77 | 79 | 74 | 78
number of drinks on peak occasion
  Baseline | 27.37 (1.98) | 25.95 (1.79) | 32.02 (1.70) | 32.15 (1.74)
  Week 4 | 22.4 (2.23) | 18.97 (2.76) | 18.18 (2.41) | 21.33 (2.32)
  Week 8 | 20.45 (2.41) | 15.85 (2.56) | 13.56 (3.15) | 17.21 (2.44)
  Week 12 | 16.80 (3.16) | 12.92 (3.18) | 12.81 (3.3) | 19.09 (2.28)
  Week 24 | 16.77 (3.36) | 13.43 (3.78) | 13.14 (3.91) | 18.01 (3.04)
  Week 36 | 13.94 (3.42) | 14.31 (3.46) | 12.46 (3.36) | 16.3 (2.73)
Statistical Analysis 1: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs XR-NTX+HRC vs Placebo+HRC; We used piecewise growth modeling to test various treatment arm effects on this outcome. Because there is currently no appropriate way to report on piecewise growth models in clinicaltrials.gov reporting tables, we are reporting the omnibus model statistics on this page called "analysis 1" and select parameters representing certain treatment arm effects on subsequent "analysis" pages. However, we note these do not constitute separate analyses, but various parameters within a single SEM model; Test type: Superiority; p = .461, Chi-squared — Denotes exact fit for the omnibus model; Complete omnibus model stats: χ2(18, N=308) = 17.93, CFI = 1.00, RMSEA < .001, SRMR = .07
Statistical Analysis 2: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs XR-NTX+HRC vs Placebo+HRC; These are select parameters for treatment arm effects that are subordinate to the omnibus model statistics in the table called "analysis 1". These are not separate analyses, but select parameters within a single SEM model. For more familiar formats, please see the related publications page, especially see https://doi.org/10.1016/s2215-0366(20)30489-2; Test type: Superiority; p = .01, z score for parameters — Linear effects of HaRT-A+XR-NTX compared to services-as usual control during treatment period; Slope = -.48, 95% CI 2-sided [-.79 to -.18] — Linear effects of HaRT-A+XR-NTX compared to services-as usual control (one of three dummy-coded variables)
Statistical Analysis 3: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs XR-NTX+HRC vs Placebo+HRC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .01, z; Slope = -.41, 95% CI 2-sided [-.67 to -.15] — Linear effects of HaRT-A+XR-NTX compared to services-as usual control (one of three dummy-coded variables) during treatment period
Statistical Analysis 4: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs XR-NTX+HRC vs Placebo+HRC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .19, z; Slope = -.23, 95% CI 2-sided [-.52 to .06] — [estimate comment as in outcome 1, analysis 3]

2. Primary Outcome: Alcohol-related Harm
Description: Using the Short Inventory of Problems, we collected data on alcohol-related harm in the past month. The range of possible scores on the single summary score is 0-45, and higher scores indicate a greater experience of alcohol-related harm.
Time Frame: Baseline, week 4, week 8, week 12, week 24, week 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | XR-NTX+HRC | Placebo+HRC | Harm-reduction Counseling (HRC) | Assessment-only
Number analyzed (Participants) | 74 | 78 | 79 | 77
score on a scale
  Baseline | 23.7 (12.03) | 23 (12.05) | 25.69 (10.25) | 22.7 (12.05)
  Week 4 | 15.33 (11.59) | 17 (11.43) | 17.98 (12.51) | 21.39 (13.67)
  Week 8 | 13.98 (12.48) | 15.52 (12.85) | 17.15 (11.97) | 18.31 (14.15)
  Week 12 | 12.15 (11.25) | 16.08 (13.2) | 15.5 (13.03) | 21 (14.06)
  Week 24 | 12.76 (12.97) | 15.89 (13.88) | 17.9 (16.19) | 16.15 (11.99)
  Week 36 | 13.35 (12.5) | 13.19 (13.4) | 16.87 (14.54) | 16.36 (13.62)
Statistical Analysis 1: Comparison: XR-NTX+HRC vs Placebo+HRC vs Harm-reduction Counseling (HRC) vs Assessment-only; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .347, Chi-squared — Denotes exact fit for the omnibus model; complete omnibus model statistics: χ2(20, N=308) = 21.89, CFI = 1.00, RMSEA = .02, SRMR = .03
Statistical Analysis 2: Comparison: XR-NTX+HRC vs Placebo+HRC vs Harm-reduction Counseling (HRC) vs Assessment-only; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .002, z — Linear effects of HaRT-A+XR-NTX compared to services-as usual control during treatment period (one of three dummy-coded variables); Slope = -2.22, 95% CI 2-sided [-3.39 to -1.06] — Linear effects of HaRT-A+XR-NTX compared to services-as usual control during treatment period (one of three dummy-coded variables)
Statistical Analysis 3: Comparison: XR-NTX+HRC vs Placebo+HRC vs Harm-reduction Counseling (HRC) vs Assessment-only; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .208, z — Linear effects of HaRT-A+placebo compared to services-as usual control during treatment period (one of three dummy-coded variables); Slope = -.82, 95% CI 2-sided [-1.89 to .25] — Linear effects of HaRT-A+placebo compared to services-as usual control during treatment period (one of three dummy-coded variables)
Statistical Analysis 4: Comparison: XR-NTX+HRC vs Placebo+HRC vs Harm-reduction Counseling (HRC) vs Assessment-only; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .025, z — Linear effects of HaRT-A only compared to services-as usual control during treatment period (one of three dummy-coded variables); Slope = -1.58, 95% CI 2-sided [-2.73 to -.42] — Linear effects of HaRT-A only compared to services-as usual control during treatment period (one of three dummy-coded variables)

3. Primary Outcome: Alcohol Frequency
Description: Addiction Severity Index (ASI - 5th edition) will be used to assess frequency of alcohol use in the past 30 days.
Time Frame: baseline, week 0, week 4, week 8, week 12, week 24, week 36
Population: see https://doi.org/10.1016/s2215-0366(20)30489-2
Measure: Mean (Standard Deviation); unit: Drinking days per month
Arm/Group | XR-NTX+HRC | Placebo+HRC | Harm-reduction Counseling (HRC) | Assessment-only
Number analyzed (Participants) | 74 | 78 | 79 | 77
Drinking days per month
  Baseline | 23.08 (7.55) | 24.63 (8.02) | 23.42 (8.63) | 23.35 (8.66)
  Week 4 | 17.87 (10.85) | 18.81 (11.45) | 17.43 (10.91) | 22.37 (10.46)
  Week 8 | 17.18 (11.83) | 18.67 (11.22) | 18 (11.8) | 20.83 (10.51)
  Week 12 | 15.15 (11.33) | 18.68 (11.45) | 15.32 (11.97) | 17.15 (10.98)
  Week 24 | 16.2 (11.82) | 18.94 (11.68) | 13.04 (11.66) | 17.93 (11.91)
  Week 36 | 15.65 (11.58) | 16.88 (11.12) | 15.02 (11.75) | 14.59 (11.51)
Statistical Analysis 1: Comparison: XR-NTX+HRC vs Placebo+HRC vs Harm-reduction Counseling (HRC) vs Assessment-only; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .028, Chi-squared — p value reflects omnibus model "close fit"; χ2(13, N=308) = 24.34, CFI = .98, RMSEA = .05, SRMR = .03
Statistical Analysis 2: Comparison: XR-NTX+HRC vs Placebo+HRC vs Harm-reduction Counseling (HRC) vs Assessment-only; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .047, z — [p-value comment as in outcome 2, analysis 2]; Slope = -4.42, 95% CI 2-sided [-8.09 to -.76] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: XR-NTX+HRC vs Placebo+HRC vs Harm-reduction Counseling (HRC) vs Assessment-only; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .009, z — [p-value comment as in outcome 2, analysis 3]; Slope = -5.95, 95% CI 2-sided [-9.72 to -2.19] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: XR-NTX+HRC vs Placebo+HRC vs Harm-reduction Counseling (HRC) vs Assessment-only; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .072, z — [p-value comment as in outcome 2, analysis 4]; Slope = -4.12, 95% CI 2-sided [-7.88 to -.36] — [estimate comment as in outcome 2, analysis 4]

4. Secondary Outcome: Motivation to Change Ruler
Description: Motivation to change will be measured using the 10-point motivation ruler, where the stem was "How motivated are you to make changes in your drinking to reduce harm?" and 1= not at all motivated and 10=totally motivated. Thus, higher scores correspond to higher motivation for alcohol harm reduction
Time Frame: baseline, week 4, week 8, week 12, week 24, week 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Assessment-only | HRC (Harm Reduction Counseling) | Placebo+HRC | XR-NTX+HRC
Number analyzed (Participants) | 77 | 79 | 78 | 73
score on a scale
  Baseline | 6.64 (2.97) | 7.49 (2.69) | 7.05 (2.94) | 6.42 (3.06)
  Week 4 | 6.37 (3) | 6.98 (3.11) | 6.43 (3.06) | 6.61 (3.02)
  Week 8 | 6.39 (3.1) | 7.48 (2.62) | 7.13 (2.79) | 6.33 (3.05)
  Week 12 | 6.08 (3.33) | 7.07 (3.14) | 6.32 (3.32) | 6.64 (3.05)
  Week 24 | 7.3 (3.07) | 6.92 (3.03) | 6.87 (3.1) | 6.59 (3.3)
  Week 36 | 7.34 (3.16) | 6.85 (3.19) | 6.71 (3.3) | 6.81 (3.07)
Statistical Analysis 1: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs Placebo+HRC vs XR-NTX+HRC; This was a mediation analysis (i.e., multiplication of regression coefficients for the regression of readiness for change slope on group (a-paths) and for the regression of alcohol outcome slopes on readiness (b-paths), where a*b is considered the mediated effect) for during-treatment effects (baseline to week 12); Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .6, z; Slope = -.12, Standard Error of Mean .24 — We used growth modeling to test mediators of the treatment effect, truncated for during-treatment effects. This analysis entails all four treatment arms; however, this specific contrast is for the XR-NTX vs control group effects on alcohol frequency
Statistical Analysis 2: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs Placebo+HRC vs XR-NTX+HRC; [analysis description as in outcome 4, analysis 1]; Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .83, z; Slope = -.04, Standard Error of Mean .18 — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs Placebo+HRC vs XR-NTX+HRC; [analysis description as in outcome 4, analysis 1]; Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .89, z; Slope = -.02, Standard Error of Mean .17 — We used growth modeling to test mediators of the treatment effect, truncated for during-treatment effects. This analysis entails all four treatment arms; however, this specific contrast is for the HaRT-A vs control group effects on alcohol frequency
Statistical Analysis 4: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs Placebo+HRC vs XR-NTX+HRC; [analysis description as in outcome 4, analysis 1]; Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .65, z; Slope = -.01, Standard Error of Mean .02 — We used growth modeling to test mediators of the treatment effect, truncated for during-treatment effects. This analysis entails all four treatment arms; however, this specific contrast is for the XR-NTX vs control group effects on alcohol quantity
Statistical Analysis 5: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs Placebo+HRC vs XR-NTX+HRC; [analysis description as in outcome 4, analysis 1]; Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .87, z; Slope = -.003, Standard Error of Mean .02 — We used growth modeling to test mediators of the treatment effect, truncated for during-treatment effects. This analysis entails all four treatment arms; however, this specific contrast is for the placebo vs control group effects on alcohol quantity
Statistical Analysis 6: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs Placebo+HRC vs XR-NTX+HRC; [analysis description as in outcome 4, analysis 1]; Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .91, z; Slope = -.002, Standard Error of Mean .02 — We used growth modeling to test mediators of the treatment effect, truncated for during-treatment effects. This analysis entails all four treatment arms; however, this specific contrast is for the HaRT-A vs control group effects on alcohol quantity
Statistical Analysis 7: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs Placebo+HRC vs XR-NTX+HRC; [analysis description as in outcome 4, analysis 1]; Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .54, z; Slope = .24, Standard Error of Mean .38 — We used growth modeling to test mediators of the treatment effect, truncated for during-treatment effects. This analysis entails all 4 treatment arms; however, this specific contrast is for the XR-NTX vs control group effects on alcohol related harm
Statistical Analysis 8: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs Placebo+HRC vs XR-NTX+HRC; [analysis description as in outcome 4, analysis 1]; Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .84, z; Slope = .06, Standard Error of Mean .32 — We used growth modeling to test mediators of the treatment effect, truncated for during-treatment effects. This analysis entails all 4 treatment arms; however, this specific contrast is for the placebo vs control effects on alcohol-related harm
Statistical Analysis 9: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs Placebo+HRC vs XR-NTX+HRC; [analysis description as in outcome 4, analysis 1]; Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .84, z; Slope = .06, Standard Error of Mean .29 — We used growth modeling to test mediators of the treatment effect, truncated for during-treatment effects. This analysis entails all 4 treatment arms; however, this specific contrast is for the HaRT-A vs control group effects on alcohol related harm

5. Secondary Outcome: Alcohol Craving
Description: Alcohol craving will be measured using the psychometrically valid, 5-item, 6-point Likert-scale Penn Alcohol Craving Scale (PACS). The score ranges from 0-30, with higher scores representing a higher level of craving.
Time Frame: baseline, week 4, week 8, week 12, week 24, week 36
Population: see https://doi.org/10.1016/s2215-0366(20)30489-2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Assessment-only | HRC (Harm Reduction Counseling) | Placebo+HRC | XR-NTX+HRC
Number analyzed (Participants) | 77 | 79 | 78 | 74
score on a scale
  Baseline | 20.74 (7.68) | 21.99 (6.18) | 21.46 (6.9) | 21.70 (5.79)
  Week 4 | 18.54 (7.15) | 17.85 (8.15) | 17.5 (9.11) | 17.19 (8.10)
  Week 8 | 16.6 (8.83) | 15.8 (8.92) | 16.15 (9.04) | 16 (8.74)
  Week 12 | 16.59 (9.77) | 14.93 (8.74) | 17.2 (8.53) | 15.25 (8.1)
  Week 24 | 15.98 (10.01) | 15.49 (8.44) | 17.09 (9.05) | 13.76 (9.13)
  Week 36 | 13.74 (9.18) | 14.87 (9.09) | 14.71 (9.09) | 14.96 (8.3)
Statistical Analysis 1: Comparison: Placebo+HRC vs XR-NTX+HRC; This was a mediation analysis (i.e., multiplication of regression coefficients for the regression of the craving (PACS) slope on group (a-paths) and for the regression of alcohol outcome slopes on readiness (b-paths), where a*b is considered the mediated effect) for during-treatment effects (baseline to week 12); Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .65, z; Slope = -.41, Standard Error of Mean .90 — We used growth modeling to test mediators of the treatment effect, truncated for during-treatment effects. This analysis entails two treatment arms: XR-NTX vs placebo effects on alcohol frequency and alcohol craving (PACS)
Statistical Analysis 2: Comparison: Placebo+HRC vs XR-NTX+HRC; This was a mediation analysis (i.e., multiplication of regression coefficients for the regression of the alcohol craving (PACS) slope on group (a-paths) and for the regression of alcohol outcome slopes on readiness (b-paths), where a*b is considered the mediated effect) for during-treatment effects (baseline to week 12); Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .46, z; Slope = -.03, Standard Error of Mean .04 — We used growth modeling to test mediators of the treatment effect, truncated for during-treatment effects. This analysis entails 2 treatment arms: XR-NTX vs placebo effects on craving and alcohol quantity
Statistical Analysis 3: Comparison: Placebo+HRC vs XR-NTX+HRC; This was a mediation analysis (i.e., multiplication of regression coefficients for the regression of alcohol craving (PACS) slope on group (a-paths) and for the regression of alcohol outcome slopes on readiness (b-paths), where a*b is considered the mediated effect) for during-treatment effects (baseline to week 12); Test type: Other — Mediation tested using the product of coefficients (a*b) approach (MacKinnon et al, 2002); p = .45, z; Slope = -.57, Standard Error of Mean .75 — We used growth modeling to test mediators of the treatment effect, truncated for during-treatment effects. This analysis entails two treatment arms: XR-NTX vs placebo effects on craving and alcohol-related harm

6. Secondary Outcome: Publicly Funded Service Utilization Costs
Description: Administrative data on publicly funded service utilization will be obtained from the King County Correctional Facility, King County Medic One/Emergency Medical Services, Harborview Medical Center (HMC), and the Washington State Comprehensive Hospital Abstract Reporting System (CHARS) for the 2-year pre-study period through the 24-week follow-up. We will obtain participant consent and HIPAA authorizations for these data at the information session. We will collect the following data: a) number of Medic One/EMS dispatches and associated costs; b) number of ER visits and associated costs; c) number of inpatient hospital admissions and total costs per admission (CHARS and HMC); d) number of bookings, length of stay and daily cost for the King County Correctional Facility. These data will be used to create overall cost outcomes.
Time Frame: 2yr pretest, 12-week treatment period, 24-week follow-up period
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | Assessment-only | HRC (Harm Reduction Counseling) | XR-NTX+HRC | Placebo+HRC
Number analyzed (Participants) | 77 | 79 | 78 | 74
US dollars
  Pretest | 722.32 (1054.45) | 829.22 (1447.25) | 583.55 (707.79) | 511.62 (665.10)
  During treatment | 1371.51 (2649.40) | 871.57 (1549.52) | 913.43 (1384.25) | 1516.09 (4274.35)
  Follow-up | 1576.97 (2871.47) | 1326.28 (2967.28) | 1286.62 (2329.87) | 1277.21 (1876.49)
Statistical Analysis 1: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs XR-NTX+HRC vs Placebo+HRC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .95, Chi-squared — Denotes exact fit for the omnibus model; Complete omnibus model : χ2(12, N=308) = .75, CFI = 1.00, RMSEA < .001, SRMR = .008
Statistical Analysis 2: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs XR-NTX+HRC vs Placebo+HRC; These are select parameters for treatment arm effects that are subordinate to the omnibus model statistics in the table called "analysis 1". These are not separate analyses, but select parameters within a single SEM model; Test type: Superiority; p = .75, Chi-squared — [p-value comment as in outcome 2, analysis 2]; Slope = -.04, 95% CI 2-sided [-.24 to .16]
Statistical Analysis 3: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs XR-NTX+HRC vs Placebo+HRC; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = .20, Chi-squared; Linear effects of HaRT-A+placebo compared to services-as usual control during treatment period (one of three dummy-coded variables); Slope = -.15, 95% CI 2-sided [-.34 to .04]
Statistical Analysis 4: Comparison: Assessment-only vs HRC (Harm Reduction Counseling) vs XR-NTX+HRC vs Placebo+HRC; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = .39, Chi-squared; Linear effects of HaRT-A compared to services-as usual control during treatment period (one of three dummy-coded variables); Slope = .10, 95% CI 2-sided [-.09 to .29]

7. Other Pre Specified Outcome: Adverse Events Due to the Study Medication
Description: The Systematic Assessment for Treatment Emergent Effects (SAFTEE) interview,68,69 which was tailored for use with this medication, includes open-ended, categorical and Likert-scale questions assessing symptoms that correspond to potential adverse events associated with XR-NTX. This measure will be embedded in the CRF and will be used to establish tolerability of the study medication. For these descriptive scores, we took the average count of adverse events reported at each time point during the study. This was a total summary score ranging from 0 to 20, where a higher score represents a higher number of adverse events experienced.
Time Frame: baseline, week 4, week 8, week 12, week 24, week 36
Measure: Mean (Standard Deviation); unit: mean scale score averaged during study
Arm/Group | XR-NTX+HRC | Placebo+HRC | Harm-reduction Counseling (HRC) | Assessment-only
Number analyzed (Participants) | 74 | 78 | 79 | 77
mean scale score averaged during study | 4.5 (3.37) | 4.88 (3.65) | 5.11 (3.38) | 4.96 (3.84)
Statistical Analysis 1: Comparison: XR-NTX+HRC vs Placebo+HRC; We conducted a generalized estimating equations analysis (negative binomial distribution, log link) to test whether number of adverse events reported increased from baseline to the follow-ups differentially across placebo and XR-NTX groups; Test type: Superiority; p > .84, z; incident rate ratio = .98, 95% CI 2-sided [.83 to 1.16]

ADVERSE EVENTS:
Time Frame: weeks 0, 4, 8, 12, 24, 36
Arm/Group | Assessment-only | HRC (Harm Reduction Counseling) | Placebo+HRC | XR-NTX+HRC
All-Cause Mortality (participants affected / at risk) | 3/77 | 0/79 | 0/78 | 0/74
Serious Adverse Events (participants affected / at risk) | 16/77 | 18/79 | 19/78 | 18/74
Other Adverse Events (participants affected / at risk) | 1/77 | 1/79 | 1/78 | 3/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assessment-only (N=77) | HRC (Harm Reduction Counseling) (N=79) | Placebo+HRC (N=78) | XR-NTX+HRC (N=74)
Hospitalization (General disorders) | 13 (13) | 17 (17) | 19 (19) | 17 (17) — One SAE was ascribed to the study procedures: difficulties ambulating due to an injection site hematoma that led to an emergency department visit, which precipitated alcohol withdrawal and subsequent hospital admission.
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
death (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — no association with procedures
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assessment-only (N=77) | HRC (Harm Reduction Counseling) (N=79) | Placebo+HRC (N=78) | XR-NTX+HRC (N=74)
Vomiting (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Event reported during study timeline that did not occur at baseline
Increased appetite (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Event reported during study timeline that did not occur at baseline
Abdominal pain (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Event reported during study timeline that did not occur at baseline
Somnolence (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Event reported during study timeline that did not occur at baseline
Decresed appetite (Product Issues) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Event reported during study timeline that did not occur at baseline
headache (Product Issues) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Event reported during study timeline that did not occur at baseline
injection site irritation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Event reported during study timeline that did not occur at baseline
dizziness (Product Issues) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Event reported during study timeline that did not occur at baseline
fatigue (Product Issues) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Event reported during study timeline that did not occur at baseline
insomnia (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Event reported during study timeline that did not occur at baseline
depressive symptoms (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Event reported during study timeline that did not occur at baseline

LIMITATIONS AND CAVEATS:
1) The treatments' relative brevity did not mirror longer-term clinical contacts this population often receives. 2) We cannot preclude experimenter bias or expectancy effects for unblinded arms. 3) Data missingness can reduce power and bias estimates, but missingness modeling lent confidence that findings are robust. 4) Generalizability may be limited by geographic location, sociodemographics, and substance-use patterns specific to the homeless population in the study area.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT01932801/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/01/NCT01932801/ICF_001.pdf